CLINICAL TRIAL: NCT06087341
Title: A Phase I Trial of Memory T Cells Expressing an NKG2D Chimeric Antigen Receptor in Children, Adolescents and Young Adults With Advanced Sarcoma
Acronym: CAR4SAR
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Antonio Pérez Martínez (Other)
Responsible Party: Sponsor-Investigator, Antonio Pérez Martínez, Chief of Pediatric Hemato-Oncology and Hematopoietic Transplantation Service, Instituto de Investigación Hospital Universitario La Paz
Organization: Instituto de Investigación Hospital Universitario La Paz (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CAR4SAR
Record Dates: First submitted 2023-10-11; First posted 2023-10-17 (Actual); Last update posted 2024-04-12 (Actual); Status verified 2024-04

CONDITIONS: Advanced Sarcoma

STUDY DESIGN:
Intervention Model Description: Arm A: systemic transduced donor-derived NKG2D-CAR memory T cells infusion. Arm B: dual treatment, with both systemic and locally transduced donor-derived NKG2D-CAR memory T cells infusion.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NKG2D-CAR memory T cells infusion (Experimental): If the primary tumor and/or metastases are not accessible, the patient will be included in Arm A.This group will receive an intravenous infusion of NKG2D-CAR memory T cells.
  Interventions: Other: NKG2D-CAR memory T cell
- Systemic and locally transduced NKG2D-CAR memory T cells infusion (Experimental): If the primary tumor and/or metastases are accessible, the patient will be included in Arm B. This group will receive an intravenous infusion of NKG2D-CAR memory T cells and an intratumoral dose of NKG2D-CAR memory T cells.
  Interventions: Other: NKG2D-CAR memory T cell

INTERVENTIONS:
Other: NKG2D-CAR memory T cell — Patients will be allocated in two groups: Arm A and Arm B. Both groups will receive an intravenous infusion of NKG2D-CAR memory T cells. Additionally, patients on Arm B will receive an intratumoral dose of NKG2D-CAR memory T cells (in accessible primary tumor and metastases). The distribution of patients on one arm or other will depend on their clinical characteristics described in the inclusion/ exclusion criteria. All patients will receive lymphodepleting chemotherapy prior to the infusion of NKG2D-CAR memory T cells according to the usual clinical practice in our center. Some patients will also receive low dose radiotherapy prior to infusion.

SUMMARY:
Phase I, open label, prospective, single-center, non-randomized, dose escalation clinical trial aiming to determine the dose-limiting toxicity (DLT) and maximum tolerated dose (MTD) of systemic transduced donor-derived NKG2D-CAR memory T cell infusions (Arm A), and of dual treatment, with both systemic and locally transduced donor-derived NKG2D-CAR memory T cell infusions (Arm B).

DETAILED DESCRIPTION:
Childhood cancer is considered a rare disease based on prevalence. Despite this, in developed countries, cancer is the most common cause of disease-related death in the pediatric population. Sarcomas are a rare and heterogeneous group of malignant tumors of mesenchymal origin representing around 10% of pediatric cancers. For patients with standard-risk and localized disease, survival is 70-80%. However, for those patients with high-risk disease, or those who relapse or develop metastases, the survival rate is only 30%. Current treatment consisting in local surgery, radiotherapy and poly-chemotherapy remains ineffective in advanced stages or relapse and is associated with acute and chronic adverse effects which compromise survival and quality of life. Thus, there is an urgent need to find new therapeutic alternatives in order to improve the outcome in sarcoma patients. Different groups have described the importance of NKG2D receptor and NKG2D ligands (NKG2DL) in sarcoma immunosurveillance. Tumor cells are recognized and eliminated by the immune surveillance system. A master key receptor called NKG2D is critical to induce cancer control. Recently, this group has published how this receptor can recognize and target most childhood cancers including sarcoma. Although different cells from the surveillance system possess this receptor, cancer cells can block their ability to recognize and eliminate the tumor cells. NKG2D CAR receptor induces tumor-specific lysis, is safe to normal cells and provides effector cells the ability to bypass the mechanisms of resistance induced by tumor cells. In the present study the investigators aim to analyze the safety of an NKG2D-CAR T cell therapy in pediatric, adolescent and young adult (AYA) patients suffering from advanced sarcoma. In a recent preclinical study developed by this group, the investigators demonstrated the efficacy and safety of an NKG2D-CAR T cell-based therapy for osteosarcoma. Furthermore, in this hospital, NKG2D-CAR T cells have been already produced in a GMP-environment and infused in two pediatric patients as compassionate use, and no signs of treatment-related toxicity have been observed. In the present study, the investigators aim to develop a dose escalation Phase I trial of NKG2D chimeric antigen receptor-T cells (NKG2D-CAR T) to assess the safety and clinical activity in pediatric patients with advanced sarcoma. This clinical trial proposal is the continuation of a previous research project funded by the Asociación Española Contra el Cáncer (AECC) in 2016, which was the first AECC funded project on CAR T cell therapy in children with metastatic disease.

ELIGIBILITY:
Inclusion Criteria:

* Age: ≤ 40 years at the time of recurrence or progression with any type of sarcoma that has recurred or not responded to standard therapy and is deemed incurable by standard therapy.
* Positive NKG2DL expression in sarcoma samples. Ideally, they should have centralized histological verification of NKG2DL expression in sarcoma samples (positive expression is defined as at least 2+ expression (0-4+ scale) in >50 percent of the tumor cells using anti-MICA and or anti-ULBP2). Patients will undergo biopsy following enrollment to obtain tissue to assess NKG2DL expression, with the following restrictions:

  * If the patient doesn´t have adequate accessible tumor for biopsy (at least 1 cm diameter).
  * Procedures employed to acquire biopsies for tumor lysates will be limited to percutaneous needle or core biopsies, thoracoscopic excision or open biopsies of readily accessible lesions. Pulmonary lesions may be biopsied but extensive surgery such as thoracotomy or laparotomy should not be employed.
  * Patients who require biopsy should not be enrolled if in the opinion of the principal investigator (PI), the tumor site places the patient at substantial related risk from the biopsy procedure.

In patients that fulfill any of these restrictions, when adequate archived tissue is available, this may be utilized to assess NKG2DL expression.

* Patient must have either measurable or evaluable tumor.
* The tumor must be accessible for intralesional administration of CAR T cells (only in ARM B).
* Life expectancy of at least 10 weeks in opinion of the principal investigator (PI).
* Lansky (age <16 years) or Karnofsky (age >=16 years) score of 50 or greater.
* Patients must have recovered from the acute toxic effects of all prior anticancer therapy (including chemotherapy and radiotherapy).
* Adequate bone marrow function defined by an absolute neutrophil count (ANC) of >/= 1.000/μL, platelet count of >/= 30.000/μL and hemoglobin of >/= 9.0 g/dl, and absence of a regular red blood cell and platelet transfusion requirement.
* Patients should have a normal hepatic function with a total bilirubin <2 times the upper limit of normal and serum glutamic oxaloacetic transaminase (SGOT) or serum glutamic pyruvic transaminase (SGPT) < 2 times the upper limit of normal, and adequate renal function as defined by a serum creatinine ≤ 1.5 upper limit of normal.
* Patient or patient's legal representative, parent(s), or guardian able to provide written informed consent.
* Sexually active patients must be willing to utilize one of the more effective birth control methods for 6 months after the infusion. Male partner should use a condom.

Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, unless they are using highly effective methods of contraception while taking study treatment and for at least 6 months after the NKG2D-CAR T infusion and until CAR-T cells are no longer present by qPCR on two consecutive tests. Highly effective contraception methods include, as defined by the CTFG recommendations (available at h t t p s : / / w w w . h m a . e u / f i l e a d m i n / d a t e i e n / H u m a n _ M e d i c i n e s / 0 1 -About_HMA/Working_Groups/CTFG/2014_09_HMA_CTFG_Contraception.pdf):

* Combined (estrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation (oral, intravaginal, transdermal)
* Progestogen-only hormonal contraception associated with inhibition of ovulation (oral, injectable, implantable)
* Intrauterine device (IUD)
* Intrauterine hormone-releasing system
* Bilateral tubal occlusion
* Vasectomised partner (provided that partner is the sole sexual partner of the trial participant and that the vasectomised partner has received medical assessment of the surgical success)
* Sexual abstinence (only if defined as refraining from heterosexual intercourse during the entire period of risk associated with the study treatments. The reliability of sexual abstinence needs to be evaluated in relation to the duration of the clinical trial and the preferred and usual lifestyle of the subject).

Sexually active males should use a condom during intercourse while taking study treatment and for at least 6 months after the infusion and until CAR-T cell are no longer present by qPCR on two consecutive tests.

Exclusion Criteria:

* Enrolled in another treatment protocol.
* Evidence of untreated and active infection or clinically significant systemic illness:

  * Cardiac disorder defined as LVFE < 45% determined by ECHO.
  * Human Immunodeficiency Virus (HIV) positive test.
  * Presence of active or prior CMV, EBV, hepatitis B or C as indicated by serology.
  * Any significant pulmonary, hepatic or other organ dysfunction.
* Chronic corticosteroid dependence (except replacement therapy).
* Evidence of any toxicity grade ≥ 4 (according to Common Terminology Criteria for Adverse Events (CTCAE) Version 5.0).
* Pregnant or lactating women.
* Medical history of epilepsy.
* Any other condition that, in the opinion if the PI, may interfere with the efficacy and/or safety evaluation of the trial.

Max Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 18 (Estimated)
Dates: Start 2024-01-10 (Actual); Primary Completion 2028-01 (Estimated); Study Completion 2028-04 (Estimated)

PRIMARY OUTCOMES:
Safety: Dose-limiting toxicity (DLT) of NKG2D-CAR memory T cells | During the study treatment, until 28 days after the last study iv treatment administration
  1. Any grade 3 or higher toxicity with an attribution of definitely or probably related to the infusion of the NKG2D CAR-T cells with the exception of Grade 3 fever and immediate hypersensitivity reactions occurring within 2hours of cell infusion that are reversible to a Grade 2 or less within 24 hours of cell administration with standard therapy;
  2. Any lower grade toxicity that increases to a grade 3 or higher as a direct result of the NKG2D CAR-T cell infusion.
Safety: Maximum Tolerated Dose (MTD) of NKG2D-CAR memory T cells | During the study treatment, until 28 days after the last study iv treatment administration
  The highest dose level if no Dose-limiting toxicitys are observed
Response rate | At day 60 after the treatment
  This outcome will be evaluated by Immune-Related Response Criteria (iRECIST) v1.1.
  The efficacy will be measured by objective response rate (ORR) at D60 in both arms, which includes Complete Response (CR) and Partial Response (PR) based on Immune-Related Response Criteria iRECIST v1.1.

SECONDARY OUTCOMES:
Rate of NKG2D-CAR T cells persistence in peripheral blood | During 12 months after the treatment
  Number of Arm A and Arm B subjects with persistence of NKG2D-CAR T cells in peripheral blood at screening and then starting from D1.
Rate of NKG2D-CAR T cells persistence in the tumor and metastasis site | 21 and 60 days after the treatment
  Number of Arm A and Arm B subjects with persistence of NKG2D-CAR T cells in the tumor samples at biopsy times (D21 and D60).
Rate of NKG2DL positive expression on primary sarcoma samples | 21 and 60 days after the treatment
  Number of Arm A and Arm B subjects with persistence of NKG2D-CAR T cells in peripheral blood at D21 and D60.
Cytokine determination in the serum of patients | During 12 months after the treatment
  Obtain primary patient-derived cancer cells from accessible sarcomas
Analysis of patient peripheral blood immune cell subpopulations | 21 and 60 days after the treatment
  Identify the immune cell phenotypes linked to CAR-T expansion and response provides an opportunity to understand the mechanisms of CAR-T success and craft approaches to improve CAR-T activity. The changes in cell differentiation stages and exhaustion markers of immune populations will be done by spectral flow cytometry.
Identify the DNA methylation profile of NKG2DL (MICA, MICB AND ULBPS 1-3) in primary sarcoma samples and DNA methylation profile of NKG2D-T cells before and after infusion. | 21 and 60 days after the treatment
  Analyze the DNA methylation profile of MICA, MICB and ULBP1-3 genes in primary sarcoma samples from D0, D21 and D60, by pyrosequencing techniques.
Evaluate the presence of soluble NKG2DL and ANTI-MICA antibodies in the serum of patients under therapy | During 60 days after the treatment
  The presence of anti-MICA antibodies will be determined in the serum of patients obtained at different times using LABScreen assay by Luminex Technology (LABScreen TM MICA and LSA-MIC single antigen, One Lambda and Diagnostica Longwood, respectively).

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitario La paz, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No